CLINICAL TRIAL: NCT06862154
Title: Femoral Nerve Block Versus Intravenous Fentanyl for Pain Management in Emergency Department Patients With Hip Fracture: A Randomized, Double-Blind, Clinical Trial
Brief Title: Comparison of the Efficiency of Femur Nerve Block and Intravenous Analgesia Treatment in Hip Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Sinan Karacabey, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09.2022.604
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures; Analgesia; Femoral Nerve
Keywords: Ultrasound guided analgesia; pain control
MeSH Terms: conditions — Hip Fractures; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind, randomized controlled design to compare ultrasound-guided femoral nerve block (FNB) and intravenous fentanyl for pain management in hip fracture patients. To maintain blinding, all patients receive two interventions: one active treatment and one placebo. The FNB group receives an active femoral nerve block (bupivacaine) and a placebo IV infusion (saline), while the IV fentanyl group receives active IV fentanyl and a placebo femoral block (saline).
  A non-blinded investigator prepares all syringes and IV bags, labeled as "Treatment A" and "Treatment B", ensuring that the patients, treating physicians, and outcome assessors remain blinded. Pain assessments and opioid use are recorded by a blinded investigator. This rigorous masking protocol minimizes bias and enhances the validity of the study's findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): Patients in this group receive an ultrasound-guided, single-injection femoral nerve block using 20 mL of 0.5% bupivacaine. This intervention aims to provide effective regional analgesia, reducing preoperative pain and opioid requirements. A placebo intravenous infusion (100 mL normal saline) is administered to maintain blinding.
  Interventions: Procedure: Femoral Nerve Block
- IV Analgesia-Fentanyl (Active Comparator): Patients in this group receive intravenous fentanyl at 1 mcg/kg, diluted in 100 mL normal saline, for systemic pain control. To ensure blinding, a placebo femoral nerve block with 20 mL of normal saline is performed. Pain scores and opioid consumption are assessed to compare the efficacy of both approaches.
  Interventions: Drug: IV Analgesia- Fentanyl

INTERVENTIONS:
Drug: IV Analgesia- Fentanyl — Patients receive intravenous fentanyl at a dose of 1 mcg/kg, diluted in 100 mL normal saline, administered as a single dose for systemic analgesia. This intervention aims to control acute pain in hip fracture patients before surgical intervention.
  Arms: IV Analgesia-Fentanyl
Procedure: Femoral Nerve Block — Patients undergo an ultrasound-guided, single-injection femoral nerve block with 20 mL of 0.5% bupivacaine. This regional anesthesia technique targets the femoral nerve, providing effective pain relief while reducing opioid requirements.
  Arms: Femoral Nerve Block

SUMMARY:
It is well-established that hip fractures impose a significant medical, socioeconomic, and financial burden. In the elderly population, the associated mortality and morbidity are particularly pronounced: within one year following a hip fracture, mortality rates range from 20% to 30%; approximately one-third of patients require an elevated level of care, and only 30-40% retain the potential to fully recover and regain their pre-injury functional status. Consequently, strategies to enhance early outcomes in these patients are urgently needed. Reducing preoperative pain has been shown to improve patient satisfaction, facilitate the timing and effectiveness of physical therapy, shorten hospital stays, and support long-term functional recovery. Perioperative nerve blockade has demonstrated superior efficacy compared to systemic analgesia, traction, neurostimulation, and alternative medicine approaches. The advantages of peripheral nerve blocks include reduced pain scores, decreased opioid consumption, a lower risk of pneumonia, shorter time to ambulation, diminished postoperative cognitive dysfunction, and a more cost-effective analgesic regimen. This study seeks to evaluate the effects of femoral nerve block (FNB) on common hip fracture types within a trauma patient population. Specifically, we compared the efficacy of ultrasound-guided, single-injection femoral nerve block against prevalent hip fracture types prior to surgery, assessing outcomes longitudinally through changes in pain scores and opioid requirements.

DETAILED DESCRIPTION:
Hip fractures constitute a significant medical and socioeconomic challenge, particularly among elderly populations. Epidemiological projections estimate a marked rise in the global incidence of hip fractures, with approximately 6.26 million cases anticipated by 2050. These injuries are associated with substantial morbidity and mortality, with one-year post-fracture mortality rates ranging from 20% to 30%. Furthermore, only 30% to 40% of survivors recover their pre-injury functional capacity, and many require long-term care, underscoring the profound impact of these injuries.

Effective pain management is pivotal in optimizing early outcomes for patients with hip fractures. Adequate analgesia not only enhances patient comfort but also facilitates the initiation of physical therapy, shortens hospital stays, and supports improved long-term functional recovery. Various pain control strategies, including systemic analgesia, traction, neurostimulation, and alternative therapies, have been employed. However, perioperative nerve blockade has demonstrated superior efficacy and broader patient benefits. Peripheral nerve blocks, such as the femoral nerve block (FNB), offer notable advantages, including reduced pain scores, decreased opioid consumption, lower incidence of pneumonia, enhanced mobilization, diminished risk of postoperative cognitive dysfunction, and reduced costs associated with analgesic regimens.

This randomized controlled trial seeks to evaluate the comparative efficacy of ultrasound-guided, single-injection femoral nerve block versus intravenous fentanyl for pain management in patients presenting with proximal femoral fractures in the emergency department. The study cohort comprises adult patients diagnosed with hip fractures-specifically femoral neck and intertrochanteric fractures-confirmed through radiological imaging. Participants will be randomly allocated to receive either an ultrasound-guided femoral nerve block with 20 mL of 0.5% bupivacaine or intravenous fentanyl at a dose of 1 mcg/kg.

Pain levels will be assessed using the standardized Numerical Rating Scale (NRS) at baseline (pre-intervention) and 20 minutes post-intervention. For patients with cognitive impairment, the Pain Assessment in Advanced Dementia (PAINAD) scale will serve as an alternative evaluation tool. Secondary outcomes include opioid consumption, patient satisfaction, length of stay in the emergency department, and adverse effects associated with each analgesic modality.

The study employs a double-blind methodology, ensuring that both participants and assessing clinicians remain unaware of treatment allocation. To maintain blinding, all participants will undergo two procedures: one active intervention and one placebo. In the intravenous fentanyl group, a placebo femoral block will be administered using 20 mL of normal saline, while in the FNB group, a placebo intravenous infusion (100 mL of normal saline) will be provided. This design minimizes bias in the assessment of efficacy and adverse effects.

The findings of this study are expected to inform the optimization of acute pain management strategies in emergency settings, potentially reducing opioid reliance, enhancing patient mobility, and improving overall clinical outcomes. By comparing these two analgesic approaches, this trial aims to identify the most effective and practical pain relief strategy for hip fracture patients prior to surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Radiologically confirmed proximal femur fracture (femoral neck or intertrochanteric fracture)
* Ability to provide informed consent or have a legal representative provide consent

Exclusion Criteria:

* Hemodynamic instability (SBP <90 mmHg, HR >120 bpm)
* Severe trauma requiring immediate surgical intervention (e.g., multiple trauma, head injury)
* Bleeding disorders or anticoagulation therapy (INR ≥2.5, platelet count <50,000/mm³)
* Known allergy to local anesthetics (bupivacaine) or opioids (fentanyl)
* Pregnancy
* Prior administration of local anesthetic blocks or systemic opioids before arrival
* Periprosthetic fractures or previous surgery on the affected hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicy available, but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Altunbas E, Kudu E, Unal E, Sanri E, Karacabey S, Gunduz OH. Femoral nerve block vs IV fentanyl for hip fracture pain in the emergency department: A randomized double-blind clinical trial. Am J Emerg Med. 2026 Jan;99:359-364. doi: 10.1016/j.ajem.2025.10.044. Epub 2025 Oct 24. PMID 41167010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited adult patients aged 18 years and older who presented to the emergency department of Marmara University Pendik Training and Research Hospital with radiologically confirmed unilateral hip fractures (femoral neck or proximal femur). Patients were enrolled between November 2022 and December 2024.
Period: Overall Study
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl
Started | 52 | 52
Completed | 52 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 78.5 [70 to 84] | 79 [75 to 86] | 79 [71 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 25 | 34 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 52 | 52 | 104
Hypertension [Count of Participants; unit: Participants] | 34 | 33 | 67
Diabetes Mellitus [Count of Participants; unit: Participants] | 19 | 26 | 45
Chronic Heart Failure [Count of Participants; unit: Participants] | 15 | 14 | 29
Chronic Kidney Disease [Count of Participants; unit: Participants] | 4 | 5 | 9
Cancer [Count of Participants; unit: Participants] | 4 | 1 | 5
Dementia/Alzheimer [Count of Participants; unit: Participants] | 8 | 7 | 15
Multiple Myeloma [Count of Participants; unit: Participants] | 0 | 3 | 3
Other Diseases [Count of Participants; unit: Participants] | 7 | 9 | 16
Systolic Blood Pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 142 [124 to 168] | 135 [120 to 154.5] | 140 [124 to 164]
Diastolic Blood Pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 79 [74 to 89] | 78 [70 to 88] | 78 [72 to 89]
Pulse Rate [Median (Inter-Quartile Range); unit: beat per minute] | 84 [72 to 90] | 85 [76 to 102] | 84 [76 to 94]
Fracture Side [Count of Participants; unit: Participants]
  Right Side | 23 | 26 | 49
  Left Side | 29 | 26 | 55
Fracture Type [Count of Participants; unit: Participants]
  Inter trochanteric fracture | 25 | 29 | 54
  Neck of femur | 25 | 20 | 45
  Proximal femur | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Change
Description: This study assesses pain score changes from baseline to 20 minutes post-intervention in hip fracture patients. For those without cognitive impairment, the Numerical Rating Scale (NRS) is used, ranging from 0 (no pain) to 10 (worst pain), with higher scores indicating worse pain. The difference in NRS scores pre- and post-intervention evaluates the efficacy of ultrasound-guided femoral nerve block versus intravenous fentanyl. For cognitively impaired patients, the Pain Assessment in Advanced Dementia (PAINAD) scale is applied, also ranging from 0 (no pain) to 10 (severe pain), where higher scores reflect worse pain. PAINAD uses behavioral indicators like breathing and facial expression for those unable to self-report. Changes in PAINAD scores are analyzed similarly to assess treatment effectiveness.
Time Frame: Baseline (pre-intervention) and 20 minutes post-intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl
Number analyzed (Participants) | 52 | 52
units on a scale | 4 [3 to 5] | 2 [2 to 3]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (such as hypotension, nausea, headache, and dizziness) were recorded throughout the procedure and during the subsequent four-hour period.
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl
Number analyzed (Participants) | 52 | 52
Participants
  Hypotension | 0 | 3
  Headache | 0 | 5
  Dizziness | 0 | 8
  Nausea | 0 | 12
  None | 52 | 24

3. Secondary Outcome: Number of Participants With Rescue Analgesic Use
Description: Following the intervention, patients were monitored for a 4-hour period to assess the need for rescue analgesia (intravenous fentanyl, tramadol, or morphine exc).
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl
Number analyzed (Participants) | 52 | 52
Participants | 11 | 32

ADVERSE EVENTS:
Time Frame: throughout the procedure and during the subsequent four-hour period
Description: Adverse events (such as hypotension, nausea, headache, and dizziness) were recorded throughout the procedure and during the subsequent four-hour period.
Arm/Group | Femoral Nerve Block | IV Analgesia-Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 3/52
Other Adverse Events (participants affected / at risk) | 0/52 | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Femoral Nerve Block (N=52) | IV Analgesia-Fentanyl (N=52)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) — Hypotension was defined as a systolic blood pressure (SBP) <90 mmHg or a ≥20% decrease from baseline systolic blood pressure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Femoral Nerve Block (N=52) | IV Analgesia-Fentanyl (N=52)
Headache (Nervous system disorders) | 0 | 5 — Headache was defined as any new-onset or worsening head pain reported by the patient during or after the intervention.
Dizziness (Nervous system disorders) | 0 | 8 — Dizziness was defined as a subjective sensation of lightheadedness, imbalance, or the feeling that the surroundings are moving or spinning, reported by the patient during or after the procedure.
Nausea (Gastrointestinal disorders) | NA | 12 — Nausea was defined as a subjective sensation of an urge to vomit, reported by the patient during or after the procedure, regardless of whether vomiting occurred

LIMITATIONS AND CAVEATS:
First, since patients' lengths of stay in the emergency department varied, we recorded the four hours after treatment for rescue analgesia. Understanding the effect of FNB on opioid consumption would have been improved by extending this period. Second, potential side effects resulting from the treatment modalities administered (e.g. nausea, leg numbness) may have compromised treatment blinding for the researchers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT06862154/Prot_SAP_000.pdf